CLINICAL TRIAL: NCT07285720
Title: Phonological Constraints on Language Development in Individuals With Williams Syndrome
Acronym: SOUNDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PI2022_843_0021
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Williams Syndrome; Language; Phonological Short-Term Memory; EEG-NIRS
Keywords: Williams syndrome; Language; Phonological Short-Term Memory; EEG-NIRS
MeSH Terms: conditions — Williams Syndrome; Language | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with Williams syndrome (Experimental)
  Interventions: Other: EEG-NIRS protocol; Other: Questionnaire
- Patients with Down syndrome (Active Comparator)
  Interventions: Other: EEG-NIRS protocol; Other: Questionnaire
- Healthy children (Sham Comparator)
  Interventions: Other: EEG-NIRS protocol; Other: Questionnaire
- Healthy adults (Active Comparator)
  Interventions: Other: EEG-NIRS protocol; Other: Questionnaire

INTERVENTIONS:
Other: EEG-NIRS protocol — Each participant will be tested individually in a quiet room at the GRAMFC (Groupe de Recherches sur l'Analyse Multimodale de la Fonction Cérébrale, INSERM-UMR1105, Université Picardie Jules Verne and CHU Amiens-Picardie). Duration of subject's participation in the study is 120 minutes
Other: Questionnaire — Each participant will be tested individually in a quiet room at the GRAMFC (Groupe de Recherches sur l'Analyse Multimodale de la Fonction Cérébrale, INSERM-UMR1105, Université Picardie Jules Verne and CHU Amiens-Picardie). Duration of subject's participation in the study is 120 minutes

SUMMARY:
Williams syndrome (WS) is a neurodevelopmental disease characterized by mild to moderate intellectual disability and an extremely heterogeneous cognitive profile. Research has outlined two main features of WS: an atypical social behavior associated with surprising language abilities, and a hyperacusis. The purpose of this project is to investigate the relationships between both these abilities, and particularly the role of the hyperacusis on language abilities. The hyperacusis would be crucial in developing language skills: the apparent strength in the verbal domain could rely on Phonological Short Term Memory (PSTM) more in individuals with WS than in typically developing individuals. In addition, the investigators will compare individuals with WS to individuals with Down syndrome (DS): DS is often associated to strong limitations in the PSTM with poor language abilities. To this end, the investigators will use a highly innovative approach including physiological assessments (EEG-NIRS protocol) and questionnaires. The performance of people with WS will be compared to those of participants with DS and TD participants of same DA and cognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

* For SW and SD: genetic diagnosis and aged between 6- and 17 years old.
* For typical participants: any child, adolescent or young adult of the same developmental or chronological age (between 6 and 17 years of age)
* adult group (between 20 and 60 years).

Exclusion Criteria:

* Autistic Associated Disorders,
* West syndrome

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
questionnaire score of patients with WS caracterisation | 2 years
  questionnaire score for cognitive profile of patients with WS caracterisation

SECONDARY OUTCOMES:
Impact of hyperacusis on questionnaire score | 2 years
  Impact of hyperacusis on questionnaire score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No